CLINICAL TRIAL: NCT03027050
Title: T-PRF Contributes to Periodontal Healing
Brief Title: T-PRF Provides Advantages on Periodontal Healing: A Split Mouth Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Taner ARABACI, Clinical Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAP-2011301
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Periodontitis; Periodontal Attachment Loss
Keywords: periodontitis; Growth factors; Periodontal healing
MeSH Terms: conditions — Periodontitis; Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Titanium-prepared platelet rich fibrine (Experimental): T-PRF was applied with open flap debridement in test group.
  Interventions: Procedure: T-PRF; Procedure: Open Flap Debridement alone
- Open Flap Debridement alone (Active Comparator): T-PRF was not applied to control groups. Only open flap debridement was applied to control groups.
  Interventions: Procedure: T-PRF; Procedure: Open Flap Debridement alone

INTERVENTIONS:
Procedure: T-PRF — Applied for treatment of periodontal bone loss.
Procedure: Open Flap Debridement alone

SUMMARY:
It was aimed to evaluate the contributions of T-PRF treatment combined with open flap debridement on biological markers in GCF and periodontal outcomes in chronic periodontitis patients. 29 patients (58 sites) with chronic periodontitis were treated either with autologous T-PRF with OFD or OFD alone. GCF growth factor levels and relative RANKL/OPG ratio at baseline and 2, 4 and 6 weeks postoperatively were analyzed, and clinical parameters such as probing depth (PD), relative attachment level (RAL) and gingival margin level (GML) at baseline and 9 months after surgery were compromised.

DETAILED DESCRIPTION:
A total of 29 medically healthy patients (12 females and 17 males; age range 28-49 years, mean±SD: 38.22±8.21) with chronic periodontitis at the outpatient Ataturk University, Department of Periodontology, Faculty of Dentistry, Erzurum, Turkey, were selected for the study. The study, conducted from November 2015 to June 2016, was planned as a randomized, double-blinded, controlled clinical trial that used a split-mouth design. This study was proved by the ethics committee of Ataturk University Faculty of Dentistry, and all patients received verbal information regarding participation and provided written informed consent for including to the study.

Bone loss characteristics of the patients were diagnosed with full-mouth radiographs and cone-beam computed tomography. This study included the patients with moderate-to-severe chronic periodontitis with a probing depth of 5 mm or deeper and horizontal bone loss (one- or two-wall shallow interproximal defects) of at least two quadrants of the jaws after Phase-I periodontal therapy. After re-evaluating the results of Phase-I therapy, patients with any of the following were excluded from the study: 1) smoking or tobacco use in any form; 2) medications known to affect periodontal treatment and blood coagulation; 3) systemic conditions known to affect periodontal status; 4) pregnancy/lactation; and 5) poor oral hygiene (plaque index [PI] >1.5) (Sillness and Loe; 1964). Patients with teeth with 3-wall intrabony defects, gingival recession, endodontic lesion, or furcation involvement were also excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP who had pocket depth ≤ 5 mm and at least two area (grouped as Control and PRF) with horizontal bone loss after initial treatment

Exclusion Criteria:

* The subjects excluded in the study had history of systemic disease, were smokers, had allergy to any drug, had need for prophylaxis of antibiotic and had taken antibiotics at least 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Level of Growth Factor | 6 weeks
  Change from baseline growth factors levels of GCF at 6 weeks were measured by periopaper

SECONDARY OUTCOMES:
relative RANKL/OPG ratio in GCF | 6 weeks
  Change in relative RANKL/OPG ratio from baseline to 6 weeks were measured by periopaper
Alteration of Clinical Attachment Level | 9 months
  Change from baseline Clinical Attachment Levels at 9 months were measured with periodontal probe.
Alteration of Periodontal Pocket Depth | 9 months
  Change from baseline Pocket Depth at 9 months were measured with periodontal probe.
Gingival Margin Level | 9 months
  Change from baseline to 9 months were measured with periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Taner Arabacı, Principal Investigator — Ataturk University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pradeep AR, Shetty SK, Garg G, Pai S. Clinical effectiveness of autologous platelet-rich plasma and Peptide-enhanced bone graft in the treatment of intrabony defects. J Periodontol. 2009 Jan;80(1):62-71. doi: 10.1902/jop.2009.080214. PMID 19228091